CLINICAL TRIAL: NCT06349616
Title: Acute and Chronic Interventions to Improve Heat Loss During Uncompensable Humid Heat Stress in Older Adults
Brief Title: Cooling Strategies for Older Adults in the Heat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, W. Larry Kenney, Professor of Kinesiology and Physiology, Penn State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: STUDY24458
Record Dates: First submitted 2024-03-19; First posted 2024-04-05 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Aging
Keywords: Aging; Thermoregulation; Heat Stress
MeSH Terms: conditions — Heat Stress Disorders

STUDY DESIGN:
Intervention Model Description: Subjects participate in 4 experiments, 2 for each treatment (folic acid supplementation and placebo). The order of treatment is random.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Folic acid supplementation (Experimental): 5 mg/day folic acid for 6-7 weeks
  Interventions: Other: Intermittent cold-water hand and forearm immersion; Other: No intermittent cold-water hand and forearm immersion
- Control (Placebo Comparator): Cellulose placebo tablet for 6-7 weeks
  Interventions: Other: Intermittent cold-water hand and forearm immersion; Other: No intermittent cold-water hand and forearm immersion

INTERVENTIONS:
Other: Intermittent cold-water hand and forearm immersion — Participants will be seated at rest in a hot and humid environment. At 2 time points in the experiment, participants will place their hands and forearms in a bucket of cold tap water for 10 minutes.
Other: No intermittent cold-water hand and forearm immersion — Participants will be seated at rest in a hot and humid environment.

SUMMARY:
The earth's climate is warming, and the number of heat waves has increased in recent years. At the same time, the number of adults over the age of 65 is growing. Humans sweat and increase blood flow to the skin to cool their body when they get hot. Older adults do not do this as well as young adults. This makes it harder to safely be in warm and/or humid conditions. It is important to learn about cooling strategies for older adults to safely be in warm and/or humid conditions.

There is compelling evidence that intermittent hand and forearm cold-water immersion effectively reduces the rise of core temperature during heat stress in older adults. However, it is still unknown if this is an effective cooling strategy for older adults. Furthermore, our laboratory has shown that folic acid supplementation improves blood flow responses in older adults. This may be beneficial to older adults during heat stress.

DETAILED DESCRIPTION:
Subjects sign an informed consent form and undergo a medical screening prior to participation. The screening includes a physical exam, anthropometry, chemical and lipid profiles.

Subjects participate in 4 experimental trials, 2 while on folic acid supplementation and 2 while on placebo. The order of treatment (folic acid supplementation or placebo) is randomized. Participants will place their hands and forearms in cold tap water intermittently for one of the two trials for each treatment. The order of the hand and forearm immersion trial is randomized for each treatment. The trials are separated by at least five days. For each experiment, core temperature, heart rate, blood pressure, skin temperature, and sweat rate are measured. Each experimental visit will last 2 hours.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 65 and older
* English proficiency

Exclusion Criteria:

* Chron's disease, diverticulitis, or similar gastrointestinal disease
* Abnormal resting exercise electrocardiogram (ECG)
* Tobacco use
* High-risk determined by the Atherosclerotic Cardiovascular Disease (CVD) Risk Factor Assessment
* Antiepileptic or antiseizure medications
* Methotrexate

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 12 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-07-21 (Actual); Study Completion 2025-07-21 (Actual)

PRIMARY OUTCOMES:
Core temperature | A slope of core temperature for each experimental aim is calculated and reported through study completion, an average of 1 year.
  Core temperature will be monitored throughout each 2 hour experimental visit.
Heart rate | A slope of heart rate for each experimental aim is calculated and reported through study completion, an average of 1 year.
  Heart rate will be monitored continuously throughout each 2 hour experimental visit.
Blood Pressure | Blood pressure for each experimental aim is recorded and reported through study completion, an average of 1 year.
  Blood pressures will be taken every 10 minutes throughout each 2 hour experimental visit.

SECONDARY OUTCOMES:
Body Mass | Baseline immediately before beginning the experimental visit and then once again at the end of the 2 hour experimental visit
  Body weight measured on a scale
Skin Temperature | Mean skin temperature for each experimental aim is calculated and reported through study completion, an average of 1 year
  Average mean skin temperature

CONTACTS AND LOCATIONS:
Overall Officials: W. Larry Kenney, Ph.D., Principal Investigator — The Pennsylvania State University
Locations (1):
- Noll Laboratory, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No